CLINICAL TRIAL: NCT02552433
Title: Complications in Post-bariatric Body Contouring Surgery; Prevalence With hands-on Treatment Regimen
Brief Title: Complications in Body Contouring Surgery
Acronym: CONTOUR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: St. Antonius Hospital (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Valerie Monpellier, MD PhD candidate, St. Antonius Hospital
Other Study IDs: R15.035
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Bariatric Surgery; Body Contouring Surgery
Keywords: nutritional deficiencies; plastic surgery; post-bariatric; protein; skin surplus
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — Bloodsamples, asessing:
  * albumin
  * hemoglobin
  * vitamin D (25-hydroxy vitamin D)
  * ferritin
  * folic acid
  * vitamin B12
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Body Contouring Surgery: All patients who undergo BCS after bariatric surgery.
  Interventions: Dietary Supplement: protein intake assessment and optimisation

INTERVENTIONS:
Dietary Supplement: protein intake assessment and optimisation

SUMMARY:
The objective of this study is to describe the wound related complication rate in post-bariatric body contouring surgery patients who are treated according to the new Dutch guideline and to asses the factors associated with a higher complication rate.

DETAILED DESCRIPTION:
In the recently published guideline of the Dutch Association of Plastic Surgeons it is advised that assessment and improvement of the nutritional status should be part of pre-operative work-up of all post-bariatric patients who undergo body contouring surgery (BCS). The assessment should consist of consultation of a dietician and measurement of the nutritional parameters associated with wound healing. It is advised to assess the following parameters:

* albumin
* hemoglobin
* vitamin D (25-hydroxy vitamin D)
* ferritin
* folic acid
* vitamin B12

Standard treatment in this study will consist of the pre-operative work-up as advised by the guideline. Participants will have a consultation with the dietician to assess (protein) intake. In addition the first blood sample, which is part of standard treatment according to the new protocol, will be obtained to assess foregoing parameters. If there are nutritional deficiencies they will be treated according to the protocol of the department of Bariatric Surgery of the treating hospital.

To evaluate the effect of the treatment of deficiencies and to be sure that there are no deficiencies present during the BCS a second blood sample will be drawn during the body contouring procedure. For study purposes this second sample will be collected in all patients, even if a deficiency was not present at the first blood sample.

The dietician will assess current intake of the patients, with special attention the protein intake. Based on guidelines on protein-intake in post-bariatric patients and after consultation of experts (Dieticians of Maastricht University) investigators decided that the aim of the minimum protein intake is 1.5 gram per kilogram bodyweight (calculated with BMI 27kg/m2) per day. The first consultation at the dietician will be eight weeks prior to surgery. Patients will be advised to start with the extra protein-intake four weeks prior to surgery and continue this until the wounds are completely healed.

Six weeks after surgery a questionnaire will be handed-out to the patients, to assess the compliance to the treatment regime.

ELIGIBILITY:
Inclusion Criteria:

* post-bariatric patient
* undergoing BCS because of skin surplus
* contouring in one of the following regions: abdomen, mammae, legs, arms, upper body or lower body.

Exclusion Criteria:

* BMI higher than 34.9 kg/m2
* weight unstable in last 12 months
* diabetes mellitus defined by currently using either oral medication or insulin
* active smoker
* using immunosuppressive drugs, e.g. corticosteroids, methotrexate
* using anti-coagulants other than acetylsalicylic acid
* coagulopathy, vasculitis, connective tissue disorder
* kidney failure (GFR<30) or liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All post-bariatric patients with a stable weight and complaints of skin surplus can be referred to the department of Plastic and Reconstructive Surgery by the department of Bariatric Surgery or the general practitioner. After reference the treating plastic surgeon will decide whether there is an indication for BCS; the type and timing of the BCS will be at the discretion of the treating plastic surgeon. If a patient is eligible for BCS and meets the inclusion criteria the treating plastic surgeon or one of the physicians or a trained staff nurse of the plastic surgery department will explain the study and hand out patient information letter. In the second preoperative consultation informed consent will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
complication rate | 30 days
  wound related complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Aebele Mink van der Molen, MD/PhD, Principal Investigator — Sint Antonius Hospital; Maarten Hoogbergen, MD/PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (3):
- Netherlands (3):
  - Catharina Hospital, Eindhoven, North Brabant
  - Sint Antonius Hospital, Nieuwegein, Utrecht
  - Rijnstate Hospital, Arnhem